CLINICAL TRIAL: NCT01963598
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study of the Safety and Efficacy of 3-month Subcutaneous REGN1033 Treatment in Patients With Sarcopenia
Brief Title: Study of the Safety and Efficacy of REGN1033 (SAR391786) in Patients With Sarcopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1033-SRC-1239
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Dosing regimen 1
  Interventions: Drug: REGN1033 (SAR391786)
- Group 2 (Experimental): Dosing regimen 2
  Interventions: Drug: REGN1033 (SAR391786); Drug: placebo
- Group 3 (Experimental): Dosing regimen 3
  Interventions: Drug: REGN1033 (SAR391786); Drug: placebo
- Group 4 (Experimental): Dosing regimen 4
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: REGN1033 (SAR391786)
  Arms: Group 1; Group 2; Group 3
Drug: placebo
  Arms: Group 2; Group 3; Group 4

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter phase 2 study of the safety and efficacy of 3-month subcutaneous (SC) REGN1033 (SAR391786) treatment in patients with sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 70 years and older (all women participating in the study must be postmenopausal)
2. Are capable, in the investigator's opinion, to complete the study per protocol and have no significant health issues or conditions
3. Ability to follow a walking program
4. Willing and able to comply with clinic visits and study-related procedures
5. Provide signed informed consent
6. Able to understand and complete study-related questionnaires

Exclusion Criteria:

1. Hospitalization or immobilization with a duration of >48 hours within the month prior to screening
2. Surgical procedure requiring general anesthesia within 1 month prior to screening, or a planned surgical procedure requiring general anesthesia within the next 6 months
3. Participate in resistance training more than 3 times per week and regular exercise consisting of an average of 30 minutes per day or more of at least moderate physical activity
4. Chronic medications introduced within 2 weeks prior to screening
5. Respiratory disease that requires oxygen treatment
6. Cancer requiring treatment currently or in the past 3 years (except primary nonmelanoma skin cancer or in situ cervical cancer)
7. Neurological conditions that are causing impaired muscle function or mobility
8. Certain cardiovascular conditions
9. Uncontrolled diabetes

The information listed above is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial and not all inclusion/ exclusion criteria are listed.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 253 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percent change in total lean body mass | day 1 to day 85
  The primary endpoint in the study is the percent change in total lean body mass measured by DEXA (dual energy X-ray absorptiometry) from baseline (day 1) to week 12 (day 85).

SECONDARY OUTCOMES:
TEAEs | day 1 to day 141
  TEAEs (Treatment emergent adverse events) from baseline (day 1) to the end of the study (day 141).
Change in appendicular lean mass | day 1 to day 141
  Changes from baseline (day 1) in appendicular lean mass by DEXA
Change in maximal leg press strength (1-RM) | day 1 to day 141
  Change from baseline in maximal leg press strength (1-repetition max)
Change in maximal chest press strength (1-RM) | day 1 to day 141
  Change from baseline in maximal chest press strength (1-repetition max)
Change in 4M gait speed | day 1 to day 141
  Change from baseline in 4-meter (4M) gait speed
Change in SPPB subscores | day 1 to day 141
  Change from baseline in SPPB (Short Physical Performance Battery) subscores
Change in distance walked in the 6MWT | day 1 to day 141
  Change from baseline in distance walked in the 6MWT (6-Minute Walk Test)
Change in regional and total fat mass by DEXA | day 1 to day 141
  Change from baseline in regional and total fat mass by DEXA
Change in hand grip strength by handheld dynamometer | day 1 to day 141
  Change from baseline in hand grip strength by handheld dynamometer
Change in unloaded and loaded stair climb power | day 1 to day 141
  Change from baseline in unloaded and loaded stair climb power

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (43):
- United States (33):
  - Anniston, Alabama
  - Phoenix, Arizona
  - El Cajon, California
  - Garden Grove, California
  - Laguna Hills, California
  - San Francisco, California
  - Walnut Creek, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Orlando, Florida
  - South Miami, Florida
  - Chicago, Illinois
  - Baton Rouge, Louisiana
  - College Park, Maryland
  - Elkridge, Maryland
  - Boston, Massachusetts
  - Edina, Minnesota
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Athens, Ohio
  - Columbus, Ohio
  - Duncansville, Pennsylvania
  - Spartanburg, South Carolina
  - Dallas, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Richmond, Virginia
- France (4):
  - Limoges
  - Montpellier
  - Saint-Etienne
  - Toulouse
- Netherlands (3):
  - Amsterdam
  - Leeuwarden
  - Noord-Brabant
- Spain (3):
  - Albacete
  - L'Hospitalet de Llobregat
  - Madrid